CLINICAL TRIAL: NCT00002037
Title: Evaluation of the Therapeutic Benefit of r-metHuIFN- Gamma in AIDS Patients With Disseminated Mycobacterium Avium-Intracellulare (MAI) Infection: A Multi-Centered Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amgen (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 062B; IFNG-8701
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-05

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Interferon-gamma, Recombinant; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Trifluridine

INTERVENTIONS:
Drug: Trifluridine

SUMMARY:
To examine the effectiveness of subcutaneous gamma interferon in reducing severity of Mycobacterium avium- intracellulare (MAI) bacillemia episodes in AIDS patients in an open-label dose-randomized multi-center pilot clinical investigation. To evaluate the safety of gamma interferon given by subcutaneous injection (SC) in the AIDS patient in the presence and absence of AZT therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Diagnosis of AIDS and persistent Mycobacterium avium- intracellulare (MAI) bacillemia.
* Life expectancy of at least 3 months.
* Baseline chest X-ray and EKG (electrocardiogram).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Known hypersensitivity to interferons or other exogenous lymphokine.
* History of cardiac abnormality or disease.
* History of hypertension.

Patients with the following are excluded:

* Known hypersensitivity to interferons or other exogenous lymphokine.
* History of cardiac abnormality or disease.
* History of hypertension.

Prior Medication:

Excluded within 4 weeks of study entry:

* Corticosteroids.
* Anti-inflammatory medication (except aspirin).
* Changes in the dose of anti-mycobacterial drugs.
* Immune agents.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Radiotherapy.

Risk Behavior:

Excluded:

* Intravenous drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15

CONTACTS AND LOCATIONS:
Locations (1):
- New York Hosp - Cornell Med Ctr, New York, New York, United States